CLINICAL TRIAL: NCT04378036
Title: The Effects of a Hippotherapy Simulator in Children With Cerebral Palsy
Brief Title: Hippotherapy Simulator in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, canangunayyazici, Research Assistant, PhD (c), Marmara University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MarHippos
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Rehabilitation; Cerebral Palsy, Spastic
Keywords: Cerebral Palsy; Hippotherapy; Postural Balance; Gait; Postural Control
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Two different treatment methods were applied to the participants (n=30). Rehabilitation programs based on individual Neurodevelopmental Therapy were applied to the participants included in the study for eight weeks (first group). In the next eight weeks, the Hippotherapy Simulator system was applied to the same participants in addition to individual Neurodevelopmental Therapy-based rehabilitation programs (study group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurodevelopmental Therapy Group (Active Comparator): The number of participants in this group is 30. All participants were included in the rehabilitation program using only the Neurodevelopmental Therapy approach for 16 sessions (8 weeks x 2 days x 45 minutes).
  Interventions: Other: Neurodevelopmental Therapy
- Hippotherapy Simulator Group (Active Comparator): The same participants were taken into a rehabilitation program in which 16 sessions (8 weeks x 2 days a week) the Hippotherapy Simulator device (30 minutes) and Neurodevelopmental Therapy (NDT) (15 minutes) (HS + NDT method) were used together.
  Interventions: Other: Neurodevelopmental Therapy; Device: Hippotherapy Simulator

INTERVENTIONS:
Other: Neurodevelopmental Therapy — The Neurodevelopmental Therapy rehabilitation program was determined according to the children's level of gross motor function, age, gender, mental state, and preferences. Neurodevelopmental Therapy program consists of the rehabilitation of muscle tone disorders, increasing sensory-perception-motor integrity, exercises to increase limb functions and body control, stretching and strengthening exercises for muscle shortness and weakness, exercises that include movements in daily life and training activities such as standing, walking, body care.
Device: Hippotherapy Simulator — Horse Riding Simulator (HRS) device was used as a hippotherapy simulator device. HRS is a device that moves forward, backward, backward-to-back, right-to-left swing and up-and-down swing in 3 dimensions, similar to the movements of a real horse, forming an 8-shaped movement on five axes. After the children sat in the saddle section, they were first taken to the warm-up speed program for 5 minutes, then to another one of the other speed levels (gradually moved to other speed levels as appropriate for the development and tolerance of children) and finally to the warm-up speed program for 5 minutes.
  Arms: Hippotherapy Simulator Group

SUMMARY:
The aim of this study was to research the effects of hippotherapy simulator in children with Cerebral Palsy. In order to evaluate its effectiveness, assessment of gross motor functions, lower extremity functions, muscle tone and spasticity, trunk control, sitting and standing balance, walking functions and functional independence were being applied.

DETAILED DESCRIPTION:
"Cerebral Palsy (CP) describes a group of permanent disorders of the development of movement and posture, causing activity limitation, that is attributed to nonprogressive disturbances that occurred in the developing fetal or infant brain." The motor disorders of CP are often accompanied by disturbances of sensation, perception, cognition, communication, and behavior, by epilepsy, and by secondary musculoskeletal problems.

CP is the most common neurodevelopmental disorder that begins in early childhood, continues for life and causes physical impairment. Damage occurring in the developing brain results in voluntary movement, postural and motor control disorders, balance problems and gait disorders.

Hippotherapy is used effectively in increasing the participation of children with CP by improving their balance, motor function, posture and mobility and improving their quality of life. Although hippotherapy has many physical, functional, emotional and social benefits for children with CP, it also has some disadvantages that limit its use in the treatment of these children. There are risks such as serious injuries caused by children being afraid of a horse, falling from a horse or kicking a horse, increased hypertonicity due to fear and stress on the horse and exposure to allergic reactions due to environmental antigens. In order to overcome these conditions and reach more patients, hippotherapy simulator systems, which have been increasing rapidly in recent years, have been developed.

Hippotherapy simulators are systems that mimic the walking and movements of a real horse. As they are a newly developed system, studies investigating their effectiveness, especially in children with CP, are very limited. The aim of this study is to research the effects of hippotherapy simulator on gross motor functions, lower extremity functions, muscle tone and spasticity, trunk control, sitting and standing balance, walking functions and functional independence in children with Cerebral Palsy.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of Spastic Cerebral Palsy
* Children aged between 5 - 18 years
* GMFCS level is I, II or III
* Independent seating
* Walking with at least 10 meters of independent, orthotic and/or auxiliary device
* Can understand simple verbal instruction
* Those with hip adductor muscle spasticity level less than 2 according to MAS
* Having bilateral passive hip abduction enough to could sit into the hippotherapy simulator device
* Voluntarily agreed to participate in the study

Exclusion Criteria:

* Those with hip dislocation
* Severe contracture or deformity to prevent the study
* Advanced scoliosis (above 20 degrees)
* Acute uncontrolled acute seizures
* Uncontrollable severe epileptic attacks
* Visual and auditory problems
* Injection of botulinum toxin in the last 6 months patients
* Underwent surgical operation such as muscle relaxation, tendon extension, and selective dorsal rhizotomy in the last 6 months

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2017-10-28 (Actual); Study Completion 2017-10-28 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Classification System (GMFSS) | Baseline
  Functional levels of participants were determined with the "Gross Motor Function Classification System" (GMFSS) before treatment. It is a system that classifies the gross motor functions of children with cerebral palsy. It classifies gross motor functions into five levels.
Change in gross motor function from baseline to week 8 to week 16 | baseline, 8th. week, 16th. week
  The gross motor functions of the participants were evaluated using Gross Motor Function Measure-88 (GMFM-88) before treatment, in the 8th week and the 16th week. It is a valid and reliable assessment tool widely used to evaluate motor functions in children with cerebral palsy. It consists of 88 items and includes 5 subsections: (A) lying and Rolling; (B) sitting; (C) crawling and kneeling; (D) standing; (E) walking, running and jumping.
Change in range of motion from baseline to week 8 to week 16 | baseline, 8th. week, 16th. week
  The range of motion of the joints in the lower extremities was measured using the universal goniometer before treatment, in the 8th week and the 16th week.
Change in spasticity from baseline to week 8 to week 16 | baseline, 8th. week, 16th. week
  Muscle spasticity of the lower limbs was evaluated with Modified Ashworth Scale (MAS) before treatment, in the 8th week and the 16th week. In the evaluations made with MAS, the muscle tone is rated between "0" and "4". "0" indicates that there is no increase in muscle tone, and "4" indicates that the affected part is rigid in flexion and extension.
Change in muscle tones of lower extremities from baseline to week 8 to week 16 | baseline, 8th. week, 16th. week
  The tone, stiffness, and flexibility of the lower limb muscles were evaluated with the Myoton®PRO Digital Palpation Device before treatment, in the 8th week and the 16th week. It is an evidence-based Class 1 device (MDD Annex IX) that evaluates the biomechanical properties of soft biological tissues non-invasively, objectively, reliably, cheaply, quickly and easily.
Change in trunk postural control from baseline to week 8 to week 16 | baseline, 8th. week, 16th. week
  The functional strength of the trunk, postural control and quality of trunk movements were evaluated with The Trunk Impairment Scale (TIS) before treatment, in the 8th week and the 16th week. TIS has been developed to evaluate the trunk of individuals with stroke and is a scale that has been adapted for use with children with cerebral palsy. TIS evaluates the body functionally in terms of strength in the sitting position. In addition, it evaluates the relationship between the body part and function by evaluating the body's static and dynamic balances and body coordination. It consists of three subsections: static, dynamic and coordination.
Change in dynamic and functional balance from baseline to week 8 to week 16. | baseline, 8th. week, 16th. week
  The dynamic and functional balances of the participants were evaluated with The Pediatric Balance Scale (PBS) before treatment, in the 8th week and the 16th week. PBS is an assessment tool adapted from the Berg Balance Scale (BDS) to evaluate children's functional balance in daily life activities. The scale consists of 14 sections and each section is scored between 0 and 4; the highest score that can be obtained from the scale is 56.
Change in dynamic balance in sitting and standing positions from baseline to week 8 to week 16 | baseline, 8th. week, 16th. week
  Pedalo® Sensamove Balance Test Pro (Holz-Hoerz Gesellschaft mit beschränkter Haftung (GmbH), Germany) Software with miniboard was used to evaluate the dynamic balance functions of the participants during their sitting, standing position at the beginning, at the 8th and at the 16th week. This device has been developed to record the movements of the user in order to learn about the balance, response time and possible imbalances of the body.
The Functional Independence Measure (WeeFIM) | baseline, 8th. week, 16th. week
  The functional independence of children in daily activities was assessed with The Functional Independence Measure (WeeFIM) initially, at week 8 and at week 16. WeeFIM consists of 6 parts: self-care, sphincter control, mobility, locomotion, communication, and social communication, and a total of 18 activities are questioned. It is scored from 1 to 7 according to whether it receives help, performs on time or whether an auxiliary device is required when performing the function in each item.
Change in walking functions from baseline to week 8 to week 16 | baseline, 8th. week, 16th. week
  Win-Track (Medicapteurs, France) path and software system was used to evaluate the walking functions (Spatio-temporal parameters) of participants at the beginning, in the 8th and the 16th week. Win-Track; static, posturography and gait analysis is a foot pressure-sensitive walking path that provides complete freedom in posture and movement acquisition. It records foot pressure up to 200 images per second during standing, walking or certain activities (such as sports movements, postural sequences) through 12.288 sensors on the Win-Track, which is in the form of a one-piece platform.

CONTACTS AND LOCATIONS:
Overall Officials: Canan GÜNAY YAZICI, PhD(c), Principal Investigator — Marmara University Institute of Health Sciences; Zübeyir SARI, Assoc Prof, Study Director — Marmara University Faculty of Health Sciences
Locations (1):
- Özdel Dilbade Özel Eğitim ve Rehabilitasyon Merkezi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Garvey MA, Giannetti ML, Alter KE, Lum PS. Cerebral palsy: new approaches to therapy. Curr Neurol Neurosci Rep. 2007 Mar;7(2):147-55. doi: 10.1007/s11910-007-0010-x. PMID 17324366
- [Background] Papavasiliou AS. Management of motor problems in cerebral palsy: a critical update for the clinician. Eur J Paediatr Neurol. 2009 Sep;13(5):387-96. doi: 10.1016/j.ejpn.2008.07.009. Epub 2008 Sep 7. PMID 18778959
- [Background] Zadnikar M, Kastrin A. Effects of hippotherapy and therapeutic horseback riding on postural control or balance in children with cerebral palsy: a meta-analysis. Dev Med Child Neurol. 2011 Aug;53(8):684-91. doi: 10.1111/j.1469-8749.2011.03951.x. Epub 2011 Mar 24. PMID 21729249
- [Background] Meregillano G. Hippotherapy. Phys Med Rehabil Clin N Am. 2004 Nov;15(4):843-54, vii. doi: 10.1016/j.pmr.2004.02.002. PMID 15458756
- [Background] Lee DR, Lee NG, Cha HJ, Yun Sung O, You SJ, Oh JH, Bang HS. The effect of robo-horseback riding therapy on spinal alignment and associated muscle size in MRI for a child with neuromuscular scoliosis: an experimenter-blind study. NeuroRehabilitation. 2011;29(1):23-7. doi: 10.3233/NRE-2011-0673. PMID 21876292
- [Background] Lee CW, Kim SG, Na SS. The effects of hippotherapy and a horse riding simulator on the balance of children with cerebral palsy. J Phys Ther Sci. 2014 Mar;26(3):423-5. doi: 10.1589/jpts.26.423. Epub 2014 Mar 25. PMID 24707098
- [Background] Palisano R, Rosenbaum P, Walter S, Russell D, Wood E, Galuppi B. Development and reliability of a system to classify gross motor function in children with cerebral palsy. Dev Med Child Neurol. 1997 Apr;39(4):214-23. doi: 10.1111/j.1469-8749.1997.tb07414.x. PMID 9183258
- [Background] Palisano RJ, Hanna SE, Rosenbaum PL, Russell DJ, Walter SD, Wood EP, Raina PS, Galuppi BE. Validation of a model of gross motor function for children with cerebral palsy. Phys Ther. 2000 Oct;80(10):974-85. PMID 11002433
- [Background] Glanzman AM, Swenson AE, Kim H. Intrarater range of motion reliability in cerebral palsy: a comparison of assessment methods. Pediatr Phys Ther. 2008 Winter;20(4):369-72. doi: 10.1097/PEP.0b013e31818b7994. PMID 19011528
- [Background] Mutlu A, Livanelioglu A, Gunel MK. Reliability of Ashworth and Modified Ashworth scales in children with spastic cerebral palsy. BMC Musculoskelet Disord. 2008 Apr 10;9:44. doi: 10.1186/1471-2474-9-44. PMID 18402701
- [Background] Schneider S, Peipsi A, Stokes M, Knicker A, Abeln V. Feasibility of monitoring muscle health in microgravity environments using Myoton technology. Med Biol Eng Comput. 2015 Jan;53(1):57-66. doi: 10.1007/s11517-014-1211-5. Epub 2014 Oct 21. PMID 25331739
- [Background] Saether R, Helbostad JL, Adde L, Jorgensen L, Vik T. Reliability and validity of the Trunk Impairment Scale in children and adolescents with cerebral palsy. Res Dev Disabil. 2013 Jul;34(7):2075-84. doi: 10.1016/j.ridd.2013.03.029. Epub 2013 May 1. PMID 23643761
- [Background] Franjoine MR, Gunther JS, Taylor MJ. Pediatric balance scale: a modified version of the berg balance scale for the school-age child with mild to moderate motor impairment. Pediatr Phys Ther. 2003 Summer;15(2):114-28. doi: 10.1097/01.PEP.0000068117.48023.18. PMID 17057441
- [Background] Kucukdeveci AA, Yavuzer G, Elhan AH, Sonel B, Tennant A. Adaptation of the Functional Independence Measure for use in Turkey. Clin Rehabil. 2001 Jun;15(3):311-9. doi: 10.1191/026921501676877265. PMID 11386402
- [Background] Kim DY, Lim CG. Effects of Pedalo(R) training on balance and fall risk in stroke patients. J Phys Ther Sci. 2017 Jul;29(7):1159-1162. doi: 10.1589/jpts.29.1159. Epub 2017 Jul 15. PMID 28744037
- [Background] Ramachandra P, Maiya AG, Kumar P. Test-retest reliability of the Win-Track platform in analyzing the gait parameters and plantar pressures during barefoot walking in healthy adults. Foot Ankle Spec. 2012 Oct;5(5):306-12. doi: 10.1177/1938640012457680. Epub 2012 Sep 5. PMID 22956663

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT04378036/Prot_SAP_ICF_000.pdf